CLINICAL TRIAL: NCT01717430
Title: Repeated Epidural and Sacroiliac Joint Glucocorticoid Injections and Their Effect on Hypothalamic-Pituitary-Adrenal Axis Suppression and Metabolic Status
Brief Title: Metabolic and Endocrine Effects of Repeated Epidural and Sacroiliac Joint Corticosteroid Injections
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Ryan Amadeo, Assistant Professor, University of Manitoba
Other Study IDs: B2012:062
Record Dates: First submitted 2012-10-08; First posted 2012-10-30 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Neck Pain; Back Pain
Keywords: Injections, epidural; Injections, intra-articular; Chronic pain; Neck pain; Back pain; Low back pain; Sciatica; Sacroiliac joint; Corticosteroids; Dexamethasone; Adrenocorticotropic hormone; Adrenal insufficiency; Hemoglobin A, glycosylated
MeSH Terms: conditions — Neck Pain; Back Pain; Chronic Pain; Low Back Pain; Sciatica; Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Corticosteroid injection: Consecutive patients receiving initial or repeated sacroiliac joint or single or multi-level epidural corticosteroid injections as part of their management plan for SI joint, neck, back, or radicular pain. Injections will be performed using 0.5 mL bupivacaine 0.25% and 15 mg dexamethasone sodium phosphate.

SUMMARY:
Corticosteroid injections into the epidural space or sacroiliac joint are increasingly used for the treatment of chronic neck, low back, and leg pain. These injections may have several side effects, including suppression of the body's adrenal glands to produce steroids (adrenal suppression) and negative effects on metabolism (weight gain, increased blood pressure, and high blood sugar levels).

The purpose of this study is to determine the time course and predictors of adrenal suppression and the metabolic effects of corticosteroid injections for chronic pain.

The investigators hypothesize normalization of adrenal function to occur within three weeks of injection in most individuals. An increased frequency of injections is predicted to lead to prolonged adrenal suppression. Corticosteroid injections are also hypothesized to lead to increases in body weight, blood pressure, and blood sugar levels, particularly in diabetic individuals.

DETAILED DESCRIPTION:
Interventional pain procedures using corticosteroid injections (CIs), such as epidural steroid injections (ESIs) and sacroiliac joint injections (SIJIs), may have adverse metabolic and endocrine effects, including suppression of the hypothalamic-pituitary-adrenal axis (HPAA), hypertension, weight gain, and hyperglycemia. Based on sparse data on these adverse effects following repeated, long-term CIs, current guidelines suggest a maximum frequency of four to six injections annually, even though patients may benefit from more frequent treatments.

This prospective cohort study will follow first-time or repeat ESI or SIJI patients receiving injections with 0.5 mL bupivacaine 0.25% and 15 mg dexamethasone sodium phosphate at a maximum frequency of once every six weeks in order to:

* determine the frequency and duration of HPAA suppression;
* determine the incidence and predictors of prolonged (≥ 3 weeks) HPAA suppression;
* determine the baseline incidence and predictors of HPAA suppression in chronic pain patients presenting for their first CI; and
* determine the effect of CIs on body weight, resting blood pressure, and glycemic control over a six-month period.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving SI joint or epidural corticosteroid injections
* At least 18 years of age

Exclusion Criteria:

* Contraindication to corticosteroid injection (infection; pregnancy; uncontrolled diabetes mellitus [per patient's report]; active congestive heart failure; coagulopathy; medical conditions that prohibit holding anticoagulant or antiplatelet therapy, with the exception of aspirin, for at least two weeks prior to injection; and allergy to iodinated contrast dye, corticosteroids, or amide local anesthetics)
* Known disorder of the hypothalamic-pituitary-adrenal axis
* Corticosteroid injection within 6 weeks of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving initial or repeated sacroiliac (SI) joint injections or single- or multi-level epidural injections with corticosteroids as part of their management plan for chronic SI joint, neck, back, or radicular pain.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2012-10; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Time to Normalization of Hypothalamic-Pituitary-Adrenal Axis (HPAA) Function Following Epidural or Sacroiliac Joint Corticosteroid Injection | From date of enrollment (Baseline) until the date of HPAA normalization assessed every 3 weeks up to 6 months
  The high-dose rapid adrenocorticotropic hormone (ACTH) stimulation test will be performed to determine if HPAA suppression is present. Serum cortisol will be measured by electrochemiluminescence immunoassay immediately prior to and at 30 and 60 min following injection of 250 mcg cosyntropin IV. A serum cortisol level <550 nmol/L (<20 mcg/dL) at either time point following cosyntropin administration will designate HPAA suppression.

SECONDARY OUTCOMES:
Incidence of Hypothalamic-Pituitary-Adrenal Axis (HPAA) Suppression in Patients Presenting for Corticosteroid Injection | Baseline
  The high-dose rapid ACTH stimulation test will be performed at Baseline to determine if HPAA suppression is present in patients presenting for corticosteroid injection.
Incidence of Prolonged (≥ 3 weeks) Hypothalamic-Pituitary-Adrenal Axis (HPAA) Suppression Following Corticosteroid Injection | From date of injection until the date of HPAA normalization assessed every 3 weeks up to 6 months
  The high-dose rapid ACTH stimulation test will be performed to determine if HPAA suppression is present.
Change in Glycosylated HbA1c (%) from Baseline to 3 months | Baseline and 3 months
  Percent glycosylated hemoglobin (HbA1c [%]) will be measured by turbidimetric inhibition immunoassay.
Change in Glycosylated HbA1c (%) from Baseline to 6 months | Baseline and 6 months
  Percent glycosylated hemoglobin (HbA1c [%]) will be measured by turbidimetric inhibition immunoassay.
Change in Systolic Blood Pressure from Baseline to 3 weeks | Baseline and 3 weeks
Change in Systolic Blood Pressure from Baseline to 6 weeks | Baseline and 6 weeks
Change in Systolic Blood Pressure from Baseline to 3 months | Baseline and 3 months
Change in Systolic Blood Pressure from Baseline to 6 months | Baseline and 6 months
Change in Diastolic Blood Pressure from Baseline to 3 weeks | Baseline and 3 weeks
Change in Diastolic Blood Pressure from Baseline to 6 weeks | Baseline and 6 weeks
Change in Diastolic Blood Pressure from Baseline to 3 months | Baseline and 3 months
Change in Diastolic Blood Pressure from Baseline to 6 months | Baseline and 6 months
Change in Body Weight from Baseline to 3 weeks | Baseline and 3 weeks
  Percent Change in Body Weight
Change in Body Weight from Baseline to 6 weeks | Baseline and 6 weeks
  Percent Change in Body Weight
Change in Body Weight from Baseline to 3 months | Baseline and 3 months
  Percent Change in Body Weight
Change in Body Weight from Baseline to 6 months | Baseline and 6 months
  Percent Change in Body Weight

OTHER OUTCOMES:
Pain Visual Analogue Scale (PVAS) | Baseline and 3, 6, 12, and 24 weeks
  11-point scale for average pain intensity over the preceding week. Completed at Baseline, at 3 weeks following any corticosteroid injection, and at weeks 6, 12, and 24.
Functional Capacity Visual Analogue Scale (FVAS) | Baseline and 3, 6, 12, and 24 weeks
  11-point scale for average functional impairment over the preceding week. Completed at Baseline, at 3 weeks following any corticosteroid injection, and at weeks 6, 12, and 24.
Brief Pain Inventory Short Form (BPI-SF) Pain Severity and Interference Scores | Baseline and 3, 6, 12, and 24 weeks
  Completed at Baseline, at 3 weeks following any corticosteroid injection, and at weeks 6, 12, and 24.
Medical Outcome Study Short Form 36 (SF-36) Health Survey Scores | Baseline and 3, 6, 12, and 24 weeks
  Completed at Baseline, at 3 weeks following any corticosteroid injection, and at weeks 6, 12, and 24.
Oswestry Disability Index (ODI) v2.0 Scores | Baseline and 3, 6, 12, and 24 weeks
  Completed at Baseline, at 3 weeks following any corticosteroid injection, and at weeks 6, 12, and 24.
North American Spine Society Patient Satisfaction Index (PSI) | Baseline and 3, 6, 12, and 24 weeks
  Completed at Baseline (for patients with previous corticosteroid injections), at 3 weeks following any corticosteroid injection, and at weeks 6, 12, and 24.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Amadeo, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada